CLINICAL TRIAL: NCT02225028
Title: Feasibility of Telephone Counseling to Increase Physical Fitness in SCI (Co-Motion Study)
Brief Title: Feasibility of Telephone Counseling to Increase Physical Fitness in SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Charles Bombardier, Professor of Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 47327-B; 290122 (Other Grant/Funding Number: Craig H. Neilsen Foundation)
Record Dates: First submitted 2014-08-15; First posted 2014-08-25 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Spinal Cord Injury
Keywords: physical activity; physical fitness; exercise program; telephone coaching; motivational counseling; stretching; fitness improvement; exercise coaching; toning; SCI; spinal cord injury; home-based; home exercise
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity Counseling (Active Comparator): Participants who are randomized to the physical activity counseling intervention group will work with a physical activity coach over the course of 6 months to come up with a physical activity program that works for each individual. Participants will have 16 phone calls and discuss goals and values, track physical activity, troubleshoot barriers, and work on keeping exercise interesting and motivating. Participants will also learn strategies for managing stress and battling unhelpful thoughts that may get in the way of activity. By the end of the intervention, the goal is to be regularly doing 150 minutes of physical activity each week. The physical activity coach will work with participants to ensure that they are increasing activity safely in order to prevent injuries.
  Interventions: Behavioral: Physical Activity Counseling
- Usual Care (No Intervention): Participants randomized to the usual care control group will receive a packet of exercise related-information at the end of the baseline assessment as well as a letter from study staff informing them of their randomization status and their test results. The letter will provide information on biological markers that are in the at-risk range, advice to seek medical advice regarding lifestyle changes such as diet and exercise and information on how to contact study staff regarding test results. We will offer to forward test results to their health care provider provided they furnish written release of information We will emphasize our interest in providing them with a follow-up assessment in 6 months.

INTERVENTIONS:
Behavioral: Physical Activity Counseling — Participants in the physical activity counseling group will be mailed a home exercise toolkit that may include an activity monitor, exercise resistance bands, and exercise DVDs made for people with paraplegia or tetraplegia.
  Arms: Physical Activity Counseling

SUMMARY:
People with spinal cord injuries (SCI) are among the least physically active groups in our society. Approximately 1 in 4 healthy young persons with spinal cord injury (SCI) does not have sufficient fitness to perform many essential activities of daily living. About 50% of people with SCI engage in no leisure time physical activity. That is, they do not wheel or walk for pleasure, don't play a sport, don't exercise at home or go to a gym. As a result of this, cardiovascular, endocrine and metabolic conditions adversely affect the health of a large segment of the SCI population. Fortunately, clinic and/or laboratory-based aerobic conditioning and circuit training studies provide compelling evidence that people with SCI can improve their cardiorespiratory fitness and by doing so can partially reverse cardiovascular disease (CVD) risk factors, enhance Quality of Life (QOL) and improve elements of subjective well-being. While intensive, clinic-based, supervised exercise programs can improve the fitness and health of persons with SCI, the value of these findings for the SCI population is limited because the vast majority of people do not have access to these specialized programs and facilities. The gap that the present study addresses is: How can we extend the benefits of increased exercise and physical activity to more people with SCI?

The goal of this study is to evaluate the feasibility of an individually tailored, home- or community-based, telephone delivered intervention that uses evidence-based behavioral and motivational counseling to increase daily physical activity and exercise.

DETAILED DESCRIPTION:
The study is a randomized controlled trial comparing a 16 session telephone intervention aiming to increase physical activity to usual care.

Participants who agree to join the study and meet all eligibility criteria will be asked to do for following things in the course of 6 months.

BASELINE ASSESSMENT (Part 1 and 2):

For all participants who meet all screening eligibility criteria, a two-part baseline assessment will be scheduled at the University of Washington Medical Center Clinical Research Center.

During Part 1 of this visit, participants will complete an interview, medical tests and receive a DXA scan. After completing Part 1 of the baseline, participants will be given an activity monitor to wear at home for up to one week.

Approximately seven days after completing Part 1 of the baseline, participants will complete Part 2. Part 2 consists of a cardiorespiratory fitness test. A healthcare monitor will be available throughout testing to help ensure safety.

POST BASELINE FOLLOW-UP:

There are 3 possible outcomes following the baseline assessment.

1. Individuals may not be eligible for the study because of a medical condition that needs treatment (for example, diabetes or hypertension).

   Individuals who qualify for the study will be randomized (like flipping a coin) to either a usual care group or the physical activity intervention group. Participants have an equal chance of ending up in either group.
2. Participants may be randomized into the usual care group and receive no physical activity coaching by telephone.
3. Participants may be randomized into the physical activity coaching intervention group. The physical activity coach will contact participants within one week to begin the 6 month intervention.

2 AND 4 MONTH ASSESSMENT (10 minutes):

All participants, regardless of group assignment, will be asked to complete telephone interviews with the research team two and four months after completing the baseline. Interviews will consist of questions regarding physical activity levels and barriers related to exercise.

6-MONTH OUTCOME ASSESSMENT (Part 1 and 2):

After six months, all participants will be asked to return to the University of Washington Medical Center Clinical Research Center to complete the 6-month outcome assessment. The 6-month outcome assessment will be identical to the baseline assessment.

During Part 1 of this visit, participants will complete an interview, medical tests and a DXA scan. After completing Part 1 of the 6-month outcome assessment, participants will be given an activity monitor to wear at home for up to one week.

Approximately seven days after completing Part 1 of the 6-month outcome assessment, participants will complete Part 2. During Part 2 of the visit, participants will undergo a cardiorespiratory fitness test. A healthcare monitor will be available throughout testing to help ensure safety.

ELIGIBILITY:
Inclusion Criteria:

* English as primary language.
* History of traumatic SCI (C6 or below/ ASIA A-D) and uses a manual wheelchair at least 50% of the time.
* Injured at least one year prior to enrollment.
* Reports less than 150 minutes per week of moderate to vigorous physical activity.
* Presence of two or more cardiometabolic risk factors:

  1. Body Mass Index (BMI) greater than 21.
  2. Fasting high density lipoprotein cholesterol (HDL) greater than or equal to 40 mg/dL.
  3. Fasting triglycerides less than or equal to 150 mg/dL.
  4. Fasting glucose greater than or equal to 100 mg/dL.
  5. Blood pressure of 120-139 (systolic) / 80-89 (diastolic).
* Physician approval to initiate physical activity program.

Exclusion Criteria:

* Body Mass Index (BMI) greater than 40.
* Medically diagnosed ischemic heart disease; unstable angina, dysrhythmia or unstable autonomic dysreflexia; recent osteoporotic fracture, tracheostomy.
* Medically diagnosed hyperlipidemia: on lipid lowering medication or detected during baseline lipid panel.
* Medically diagnosed hypertension: on antihypertensive medication or hyertension detected during secondary screening/baseline exam.
* Engaged in a structured exercise program within 6 month of enrollment.
* Engaged in a structured diet program.
* Presence of conditions that would preclude participation in home-physical activity program such as: pressure ulcer, current substance dependence, psychosis, severe chronic upper extremity pain, surgery pending within 6 months, current infection or illness requiring hospitalization, or participation in another research study.
* Electrocardiographic abnormalities detected during any exercise test: 2o or 3o AV block, pre-excitation arrhythmia, hemi-blocks, S-T segment depression (horizontal, down sloping, or up sloping) diagnostic of myocardial ischemia, or other restrictions (ACSM Guidelines 7th Edition).
* Current use of the following medications: Lipid lowering agents (e.g., statins, fibric acid derivatives, niacins, bile-acid sequestrates, or cholesterol uptake blockers), antihyperglycemics (biguanides, sulfonyureas, incretins, TZDs), herbal medicines and hyper-vitamins having antilipemic or antihyperglycemic properties, antihypertensives (Carbonic Anhydrase Inhibitors, thiazides, or loop diuretics), and estrogen replacement therapy.
* Anticipated reasons subjects may be discharged from the trial and/or referred for medical therapy (if indicated): At the 6 month assessment subject laboratory values indicate they require medical treatment for diabetes, hyperlipidemia or hypertension; pregnancy; pressure ulcer that affects the safety of performing physical activity. NCEP ATP Guidelines will serve as the criterion for need for lipid intervention, ADA guidelines for diabetes, and JNC VII Guidelines for Hypertension

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The rate of enrollment | 1.5 years
  The investigators will measure the enrollment rate as it pertains to the feasibility of the study procedures.

SECONDARY OUTCOMES:
Study completion rate as it pertains to the feasibility of the study procedures | 6 months post randomization
  Study completion rate will be defined as participants who have not dropped out by the end of the trial and who complete the cardiorespiratory fitness test at 6 months post randomization.
Call completion rate as it pertains to the feasibility of the study procedures | 6 months post randomization
  Call completion rate will be defined as calls that lasted as least 5 minutes and addressed at least one of the planned topics during the 16 week intervention. Duration of calls will be measured by length of audio recording or coach self-report if recording is not available. Whether at least one topic was covered will be measured by audio recording review or topic completion checklist recorded by the physical activity coach.
Number of Participants with Serious and Non-Serious Adverse Events | 1.5 years
  During each intervention session the physical activity coach will ask participants whether they experienced any injuries or harm from the physical activities they performed as a part of the study. Adverse events will be recorded by the coach on a session log and discussed in a weekly supervision meeting with the study team. Serious adverse events, that is injuries or other harm related to study activities that resulted in hospitalization, will be reported to the Human Subjects board within 24 hours. The study team will discuss any serious adverse event during weekly meetings.
Missing data rates as it pertains to the feasibility of the study procedures | 1.5 years
  The data manager will run data checking programs to detect missing data fields. The target is less than 5% missing data overall among study completers.
Cardiorespiratory Fitness (V02 Peak) | Baseline and 6 months post randomization
  Cardiorespiratory fitness is defined as peak oxygen consupmtion (V02 peak) measured with open-circuit spirometry during an incremental exercise test on an arm crank ergometer. An initial workload of 10 Watts (tetraplegics) or 20 Watts (paraplegics) will be increased by 10 or 20 Watts, respectively every 3 minutes until volitional exhaustion is reached. Expired gases will be continuously analyzed by an open circuit indirect calorimetry system.
Minutes of moderate to vigorous physical activity as measured by the Physical Activity Recall Assessment for People with SCI (PARA-SCI) | Baseline and 6 months post randomization
  The PARA-SCI is a validated self-report measure of physical activity designed for people with spinal cord injuries.
Insulin Sensitivity Index (ISI) as a cardiometabolic risk factor | Baseline and 6 months post randomization
  In this test, a person fasts overnight (at least 8 but not more than 16 hours). A fasting baseline (0 minutes) blood sample (plasma glucose and insulin) will be drawn. The subject will then drink a Trutol beverage (75 grams of glucose). A second blood sample will be drawn after 2 hours (120 minutes) of Trutol consumption.
Total cholesterol to high density lipoprotein (TC:HDL) ratio as a cardiometabolic risk factor | Baseline and 6 months post randomization
  From a standard blood draw, the TC:HDL ratio will be calculated as a cardiometabolic risk factor.
Low density lipoprotein to high density lipoprotein (LDL:HDL) ratio as a cardiometabolic risk factor | Baseline and 6 months post randomization
  In a standard blood draw the LDL:HDL ratio will be calculated as a cardiometabolic risk factor.
Body Mass Index (BMI) | Baseline and 6 months post randomization
  The BMI will be calculated using height and weight during the 6 month outcome assessment.
Waist Circumference | Baseline and 6 months post randomization
  Waist circumference will be measured by research staff during the 6 month outcome assessment with a standard measuring tape.
Fat and lean body mass by dual energy x-ray absorotiometry (DXA) | Baseline and 6 months post randomization
  The procedure consists of the subject lying down on the machine for about 6-12 minutes with a low dose x-ray. The procedure is totally painless. The subject breathes normally but should remain still. The radiation is lower than a cross-country flight. Subjects should wear clothing with no metal, zippers, or buttons. All jewelry should be removed. DXA scans use a very low level of x-ray consisting of two different beams. One is a higher energy beam, while the other is a lower intensity. The lower intensity beam is only absorbed by soft tissue (muscle and fat), where as the higher intensity beam gets absorbed both by bones and by soft tissue. These differences in absorption are used to determine bone mineral density (BMD) and body composition values.

OTHER OUTCOMES:
Participant-reported changes in Pain | Baseline and 6 months post randomization
  Participants will complete self-report measures regarding pain in an interview format with the research team.
Participant-reported changes in Quality of Life | Baseline and 6 months post randomization
  Participants will complete self-report measures regarding quality of life in an interview format with the research team.

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Bombardier, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided